CLINICAL TRIAL: NCT07081035
Title: A Prospective Study Evaluating the Safety and Efficacy of Lower-Intensity INR Target (1.5-2.0) Versus Standard INR Target (2.0-3.0) in Patients Implanted With a HeartMate 3 Left Ventricular Assist Device (LVAD)
Brief Title: Trial of Low-intensity Anticoagulation to Reduce GI or Other Bleeding Complications With Equivalent Therapeutic Efficacy in HeartMate 3 LVAD Patients
Acronym: TARGET
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Min-Seok Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AMC_2025_2573
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Advanced Heart Failure; Left Ventricular Assist Devices; Anticoagulation Treatment; Bleeding Complications; Thrombotic Complications
Keywords: HeartMate 3 LVAD; Left Ventricular Assist Device; Advanced Heart Failure; Anticoagulation; Warfarin; International Normalized Ratio (INR); Low-intensity Anticoagulation; Major Bleeding; Gastrointestinal Bleeding; Pump Thrombosis; Stroke; Thromboembolism; Hemocompatibility; Randomized Controlled Trial; Safety and Efficacy
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Stroke; Thromboembolism | interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-intensity INR group (Experimental): Intervention: Drug: Warfarin (INR 1.5-2.0)
  Interventions: Drug: Warfarin (low-intensity anticoagulation)
- Standard INR group (Active Comparator): Intervention: Drug: Warfarin (INR 2.0-3.0)
  Interventions: Drug: Warfarin (standard anticoagulation)

INTERVENTIONS:
Drug: Warfarin (low-intensity anticoagulation) — Low-intensity INR group (Experimental):
  Participants will receive anticoagulation therapy with warfarin, aiming for a reduced INR range of 1.5-2.0, which is lower than the current standard recommendation. Warfarin dosing will be regularly adjusted based on INR monitoring throughout the 6-month study period.
  Arms: Low-intensity INR group
Drug: Warfarin (standard anticoagulation) — Standard INR group (Active Comparator):
  Participants will receive anticoagulation therapy with warfarin, maintaining an INR within the standard therapeutic range of 2.0-3.0. Warfarin dosing adjustments will be made regularly according to standard clinical practice and INR monitoring throughout the 6-month study period.
  Arms: Standard INR group

SUMMARY:
The TARGET trial is a prospective, single-center, randomized, open-label, active-controlled inequality clinical trial designed to evaluate the safety and efficacy of low-intensity anticoagulation therapy (target INR 1.5-2.0) compared to standard anticoagulation therapy (target INR 2.0-3.0) in patients receiving a HeartMate 3 Left Ventricular Assist Device (LVAD).

Despite the demonstrated effectiveness of HeartMate 3 LVAD in reducing thromboembolic complications, standard anticoagulation treatment guidelines recommend maintaining an INR between 2.0 and 3.0, which can lead to a substantial risk of bleeding, especially gastrointestinal (GI) bleeding. Preliminary studies, such as MAGENTUM 1, have indicated potential safety and reduced bleeding events at lower INR targets (1.5-1.9). However, robust evidence through randomized controlled trials is still required.

The primary objective of the TARGET trial is to determine if low-intensity anticoagulation therapy significantly reduces the incidence of major bleeding and thrombotic events compared to standard therapy within 6 months post-randomization. Secondary objectives include evaluating the safety and hematological complications associated with low-intensity anticoagulation.

The study will enroll adult patients aged ≥19 years who have been stably maintained on standard INR therapy (2.0-3.0) for at least 30 days post-HeartMate 3 LVAD implantation. Participants will be randomized in a 1:1 ratio into two groups: the low-intensity INR group (target INR 1.5-2.0) and the standard INR group (target INR 2.0-3.0). Randomization will be stratified based on the presence of atrial fibrillation.

The primary endpoint is a composite of hemocompatibility-related events, including major bleeding, stroke, and pump thrombosis, occurring within 6 months after randomization, as defined by INTERMACS criteria. Secondary endpoints encompass clinical outcomes such as all-cause mortality, cardiac death, LVAD-related thromboembolic events, stroke, systemic embolism, myocardial infarction, major bleeding incidents, and the rate and number of LVAD-related hospital readmissions and reoperations. Additionally, INR management outcomes, including time in therapeutic range (TTR) and frequency of warfarin dose adjustments, will be assessed.

The trial duration is approximately 36 months, including a 24-month enrollment period, a 6-month follow-up period for each participant, and time allocated for data analysis and reporting. Safety will be rigorously monitored by a Data Safety Monitoring Board (DSMB) and Clinical Events Committee (CEC), ensuring participant safety and data integrity throughout the study.

This trial aims to provide critical insights that could optimize anticoagulation strategies in LVAD patients, potentially improving patient safety by reducing bleeding risks without compromising thrombotic event protection.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet all of the following criteria will be eligible for randomization:

Adults aged ≥19 years who have successfully undergone implantation of a HeartMate 3 LVAD.

Patients who are at least 30 days post-implantation of HeartMate 3 LVAD.

Patients who have maintained stable anticoagulation therapy with standard INR (2.0-3.0) for at least 30 days post-LVAD implantation.

Patients or their legal representatives who provide documented informed consent and agree to the study protocol and follow-up schedule.

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded:

Patients implanted with any mechanical assist device other than HeartMate 3 LVAD (e.g., other LVAD models, RVAD, BiVAD).

Patients with a clinically significant stroke or transient ischemic attack (TIA) within the past 6 months.

Patients with a history of hemorrhagic stroke.

Patients who experienced major bleeding events within the past 6 months (based on INTERMACS major bleeding criteria).

Patients with uncontrolled severe hypertension (systolic ≥180 mmHg or diastolic ≥110 mmHg).

Patients requiring active treatment or surgical intervention for acute LVAD-related thrombosis or hemodynamic instability, or patients who underwent LVAD-related reoperation within the past 30 days.

Patients with severe renal dysfunction (estimated Glomerular Filtration Rate <15 mL/min) or patients undergoing dialysis.

Patients with severe liver dysfunction causing coagulation abnormalities or those classified as Child-Pugh class B or C.

Patients with active bleeding or ongoing hemorrhagic conditions.

Patients with a high bleeding risk due to:

Gastrointestinal bleeding or ulcers within the past 6 months.

Surgery involving the brain, spine, or eyes within the past 6 months.

Major central nervous system, ophthalmologic, or major open surgical procedures within the past 6 months.

Presence or suspicion of esophageal varices.

Arteriovenous malformation or vascular aneurysm.

Patients who have received thrombolytic therapy for bleeding or thromboembolism within the past 30 days.

Patients receiving long-term concurrent treatment with other anticoagulants (low molecular weight heparin, NOAC, Fondaparinux, etc.). However, temporary administration for warfarin bridging or heparin use for central venous or arterial catheter maintenance is permitted.

Patients with persistent anemia (hemoglobin <8 g/dL) or thrombocytopenia (platelet count <50,000/µL) within the past 6 months.

Patients currently experiencing infective endocarditis.

Patients with a history of severe allergy or hypersensitivity to warfarin or other anticoagulants used in this study.

Pregnant or lactating women, or women planning pregnancy during the study period.

Patients with severe terminal illness with a life expectancy of less than 12 months.

Patients with alcohol dependence or severe psychiatric conditions hindering study participation.

Patients unwilling or unable to adhere to the procedures or evaluations required by the study protocol.

Patients currently participating in another randomized drug or medical device clinical trial who have not yet completed the primary endpoint assessment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of composite hemocompatibility-related events | Within 6 months after randomization
  The primary outcome is defined as a composite of hemocompatibility-related events including major bleeding (INTERMACS major bleeding criteria), stroke (ischemic or hemorrhagic), and pump thrombosis occurring within 6 months post-randomization. Events will be centrally adjudicated based on standardized INTERMACS definitions.

SECONDARY OUTCOMES:
All-cause mortality | Within 6 months after randomization
  Incidence of death due to any cause.
Cardiac death | Within 6 months after randomization
  Incidence of death directly attributed to cardiac causes, including heart failure, myocardial infarction, or sudden cardiac death.
LVAD pump thrombosis | Within 6 months after randomization
  Incidence of pump thrombosis as defined by INTERMACS criteria, requiring intervention, replacement, or explantation of the LVAD.
LVAD-related thromboembolism | Within 6 months after randomization
  Incidence of thromboembolic events directly related to LVAD, including embolic strokes or systemic embolisms.
Transient ischemic attack (TIA) | Within 6 months after randomization
  Incidence of transient neurologic deficits lasting less than 24 hours without evidence of acute infarction.
Stroke | Within 6 months after randomization
  Incidence of ischemic or hemorrhagic stroke with clinical neurologic deficits lasting ≥24 hours, as defined by NeuroARC criteria.
Systemic embolism | Within 6 months after randomization
  Incidence of acute systemic embolism affecting major organs or limbs, confirmed by imaging or surgical findings.
Myocardial infarction | Within 6 months after randomization
  Incidence of myocardial infarction diagnosed by typical symptoms, ECG changes, and elevation of cardiac biomarkers.
Major bleeding event | Within 6 months after randomization
  Incidence of major bleeding as defined by INTERMACS major bleeding criteria, including events requiring transfusion or intervention.
Composite (cardiac death, pump thrombosis, thromboembolism) | Within 6 months after randomization
  Combined incidence of cardiac death, LVAD pump thrombosis, and LVAD-related thromboembolic events.
Composite (cardiac death, thrombosis, stroke, embolism, MI) | Within 6 months after randomization
  Combined incidence of cardiac death, LVAD pump thrombosis, stroke, systemic embolism, and myocardial infarction.
Composite (stroke, embolism, TIA, MI) | Within 6 months after randomization
  Combined incidence of stroke, systemic embolism, transient ischemic attack, and myocardial infarction.
Composite (death, stroke, embolism, TIA, MI) | Within 6 months after randomization
  Combined incidence of all-cause mortality, stroke, systemic embolism, transient ischemic attack, and myocardial infarction.
LVAD-related readmission | Within 6 months after randomization
  Incidence and frequency of hospital readmissions directly related to LVAD management or complications.
LVAD-related reoperation | Within 6 months after randomization
  Incidence and frequency of surgical reoperations directly related to LVAD complications or device malfunction.
Time in therapeutic range (TTR) | Within 6 months after randomization
  Proportion of time patients' INR values remain within the predefined therapeutic target range.
Out-of-range INR proportion | Within 6 months after randomization
  Proportion of INR measurements falling outside the predefined therapeutic target range.
Warfarin dose adjustments | Within 6 months after randomization
  Number of warfarin dose adjustments required to maintain target INR range.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Netuka I, Ivak P, Tucanova Z, Gregor S, Szarszoi O, Sood P, Crandall D, Rimsans J, Connors JM, Mehra MR. Evaluation of low-intensity anti-coagulation with a fully magnetically levitated centrifugal-flow circulatory pump-the MAGENTUM 1 study. J Heart Lung Transplant. 2018 May;37(5):579-586. doi: 10.1016/j.healun.2018.03.002. Epub 2018 Apr 11. PMID 29655662
- [Background] Rogers JG, Pagani FD, Tatooles AJ, Bhat G, Slaughter MS, Birks EJ, Boyce SW, Najjar SS, Jeevanandam V, Anderson AS, Gregoric ID, Mallidi H, Leadley K, Aaronson KD, Frazier OH, Milano CA. Intrapericardial Left Ventricular Assist Device for Advanced Heart Failure. N Engl J Med. 2017 Feb 2;376(5):451-460. doi: 10.1056/NEJMoa1602954. PMID 28146651
- [Background] Desai SR, Hwang NC. 2023 ISHLT Guidelines for Mechanical Circulatory Support. J Cardiothorac Vasc Anesth. 2023 Dec;37(12):2419-2422. doi: 10.1053/j.jvca.2023.07.044. Epub 2023 Aug 8. No abstract available. PMID 37659882
- [Background] Mehra MR, Naka Y, Uriel N, Goldstein DJ, Cleveland JC Jr, Colombo PC, Walsh MN, Milano CA, Patel CB, Jorde UP, Pagani FD, Aaronson KD, Dean DA, McCants K, Itoh A, Ewald GA, Horstmanshof D, Long JW, Salerno C; MOMENTUM 3 Investigators. A Fully Magnetically Levitated Circulatory Pump for Advanced Heart Failure. N Engl J Med. 2017 Feb 2;376(5):440-450. doi: 10.1056/NEJMoa1610426. Epub 2016 Nov 16. PMID 27959709
- [Background] Mehra MR, Goldstein DJ, Uriel N, Cleveland JC Jr, Yuzefpolskaya M, Salerno C, Walsh MN, Milano CA, Patel CB, Ewald GA, Itoh A, Dean D, Krishnamoorthy A, Cotts WG, Tatooles AJ, Jorde UP, Bruckner BA, Estep JD, Jeevanandam V, Sayer G, Horstmanshof D, Long JW, Gulati S, Skipper ER, O'Connell JB, Heatley G, Sood P, Naka Y; MOMENTUM 3 Investigators. Two-Year Outcomes with a Magnetically Levitated Cardiac Pump in Heart Failure. N Engl J Med. 2018 Apr 12;378(15):1386-1395. doi: 10.1056/NEJMoa1800866. Epub 2018 Mar 11. PMID 29526139